CLINICAL TRIAL: NCT06986447
Title: MASH/MetALD Consortium for the Assessment of Non-Invasive Testing in Monitoring Interventions, Treatment Response, and Major Liver-Related Outcomes
Brief Title: Assessment of Non-Invasive Testing in Major Liver-Related Outcomes
Acronym: MAIL-NIT
Status: Not yet recruiting | Type: Observational
Sponsor: HRI-MAIL-NIT (Industry)
Responsible Party: Sponsor
Organization: Houston Research Institute (Industry)
Other Study IDs: MAIL-NIT
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; MASLD; MASLD - Metabolic Dysfunction-Associated Steatotic Liver Disease; MASLD/MASH (Metabolic Dysfunction-Associated Steatotic Liver Disease / Metabolic Dysfunction-Associated Steatohepatitis); MetALD
Keywords: MASLD; MetALD; Non-invasive testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum and plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MASLD (Cohort A): Patients with metabolic dysfunction-associated steatotic liver disease
- MetALD (Cohort B): Patients with metabolic dysfunction-associated steatotic liver disease and increased alcohol intake

SUMMARY:
This is a general clinical research protocol to study the clinical evaluation, investigation and long-term follow up of patients who have Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) and MetALD (MASLD and increased alcohol intake), and to assess the usefulness and accuracy of non-invasive testing such as MRI and Fibroscan in tracking the progression of disease. The protocol is designed to follow the natural history, pathogenesis, interventions, treatment response, comorbidities, major liver related outcomes, and major cardiac events in patients with MASLD and MetALD, especially those with significant and advanced fibrosis. Data will be collected to help further the understanding of non-invasive testing with the hopes of lessening the need for liver biopsies in phase 3 clinical trials of MASLD and in clinical practice. Additionally, the study will aim to define the natural history of MetALD, an area that is poorly understood.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

1. Adults, 18-80, male or female.
2. Cohort A (MASH): Evidence of MASH (metabolic dysfunction-associated steatohepatitis) with fibrosis stage 3 or higher based on MRE stiffness of >3.63 kPa or liver biopsy.

   Cohort B (MetALD): Evidence of MetALD/ALD as defined by the AASLD nomenclature criteria and evidence of liver stiffness of 12 kPa or higher on VCTE.
3. Willingness to participate in the study. Exclusion criteria

<!-- -->

1. Involvement in the planning and/or conduct of the study (including sponsors, clinic staff, and vendors)
2. Participation in another clinical study with intake of an investigational product during the last 60 days prior to Baseline
3. Participation in a large multinational observational cohort (local registry and biobank are allowed) Target disease exclusions
4. History of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to baseline (For Cohort A only).
5. MELD score ≥12, as determined at baseline, due to liver disease.
6. Evidence of current, chronic liver diseases at the time of baseline:

   a. Primary biliary cholangitis b. Primary sclerosing cholangitis c. Chronic hepatitis B or D d. Hepatitis C, as defined by the presence of hepatitis C virus antibody (anti-HCV) with detected circulating ribonucleic acid (RNA) within two years prior to Screening, or during Screening Period.

   e. HCV eradication by antiviral treatment less than three years prior to Screening.

   f. History or evidence of current active autoimmune hepatitis g. History or evidence of Wilson's disease h. History or evidence of alpha-1-antitrypsin deficiency i. Evidence of genetic hemochromatosis (hereditary, primary) j. Evidence of drug-induced liver disease k. Known bile duct obstruction. l. Suspected or proven hepatocarcinoma, or metastatic tumor in the liver
7. Evidence of hepatic impairment or decompensation within 3 months prior to baseline, as defined by any of the following parameters:

   a. History of ascites, or hepatic encephalopathy b. History of variceal bleeding c. Serum albumin < 3.5 g/dL, except as explained by non-hepatic causes. d. International Normalized Ratio (INR) ≥ 1.3, except for participants under anticoagulant treatment.

   o NOTE: INR may be repeated once to reassess eligibility e. Total bilirubin (TBL) ≥ 1.5 ULN

   o NOTE: Patients with Gilbert's Syndrome are eligible with a total bilirubin above 1.5 × ULN if reticulocyte count is within normal limits (typically 0.5% to 2.5%), hemoglobin is within normal limits (typically 13.5 to 17.5 g/dL for men or 12.0 to 15.5 g/dL for women), and direct bilirubin is <20% of total bilirubin f. Platelet count < 110,000/mm3
8. Prior history of medium or large varices
9. Bariatric surgery of any kind within 2 years prior to the baseline visit Medical History and Concurrent Disease Exclusions Cardiovascular diseases
10. Any of the following diseases or procedures within 24 weeks prior to baseline:

    1. Myocardial infarction (MI)
    2. Cardiac revascularization surgery (coronary artery bypass graft / percutaneous transluminal coronary angioplasty (CABG / PTCA))
    3. Unstable angina
    4. Transient ischemic attack, stroke or cerebrovascular disease Hematological and oncological diseases
11. Active malignancy with a complete remission date within 2 years prior to the baseline visit (except for treated basal cell carcinoma or treated squamous cell carcinoma of the skin or resected carcinoma of the cervix) Other exclusion conditions
12. Immunocompromised participants such as participants that underwent organ transplantation or are diagnosed with human immunodeficiency virus (HIV) or participants with ongoing chemotherapy for stable malignant disease (such as a PD-1 inhibitor)
13. Any other known serious disease (such as major infection, clinically significant gastrointestinal disorder, major autoimmune disease) or other disease which in the Investigator's opinion would exclude the participant from the study.
14. Mental handicap, limited capacity of recognition, inability to follow the study procedures as evaluated by the Investigator, or any history of clinically important emotional and/or psychiatric illness.
15. Use of non-permitted concomitant medication within 8 weeks prior to the initial baseline visit (A transient intake < 4 weeks may be allowed after approval of the Medical Monitor)

    1. Vitamin E >400 units per day. Participants on stable vitamin E therapy (same doses) for the last 12 weeks prior to baseline are eligible but the therapy should be maintained at stable dose throughout the study
    2. Pioglitazone >15 mg per day. Participants on stable pioglitazone therapy (same doses) for the last 12 weeks prior to baseline are eligible but the therapy should be maintained at stable dose throughout the study
    3. GLP1-RA, SGLT2-I unless on stable doses for the last 12 weeks prior to baseline
    4. Amiodarone within 12 months of enrollment
    5. Methotrexate within 12 months of enrollment
    6. Chronic use (> 2 consecutive weeks) of corticosteroids with a systemic effect at doses ≥ 5 mg/day of oral prednisone (or equivalent)
    7. Tamoxifen within 12 months of enrollment
    8. Estrogens at doses greater than those used for hormone replacement or contraception
    9. Anabolic steroids except testosterone replacement
    10. Valproic acid
    11. Any other medications known to affect liver function/steatosis at the Investigator's discretion (including vitamins, herbal and dietary supplements)
16. Contraindications to MRI, including:

    1. Participants with incompatible pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field
    2. History of extreme claustrophobia
    3. The participant cannot fit inside the magnetic resonance scanner cavity

       Exclusion Criteria:

       -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be recruited solely from the clinical practices of the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 1689 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major adverse liver outcomes (MALO) | 2 years
  Variceal bleeding, hepatic encephalopathy, ascites, progression from MELD 13 to 15, liver transplant, death attributable to liver disease, progression to large varices

SECONDARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 2 years
  Fatal or non-fatal MI, fatal or non-fatal stroke, death attributable to cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Noureddin, MD, MHSc, Principal Investigator — Houston Research Institute

IPD SHARING:
Plan to Share IPD: Undecided